CLINICAL TRIAL: NCT02737709
Title: A Clinical Experience Trial to Detect the Plasma Paclitaxel Drug Concentration in Chinese Non -Small Cell Lung Cancer (NSCLC) Patients Treated With a Paclitaxel Plus Carboplatin (TC) Regimens, and Explore Individualized Treatment Using Pharmacokinetically-guided Dosing Strategy
Brief Title: Paclitaxel Detection in NSCLC Treated With TC Regimen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study have difficulty in recruiting subjectes
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, MD, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-703
Record Dates: First submitted 2016-03-22; First posted 2016-04-14 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel and Carboplatin regimen (Experimental): Paclitaxel: 175mg/m2, d1; Intravenous drip injection with 500ml N.S Carboplatin: AUC=5, d1; Intravenous drip injection with 500ml G.S Paclitaxel injection at first, followed with Carboplatin injection. 21 days per cycle; 6 cycles in total.
  Interventions: Drug: Paclitaxel and Carboplatin regimen

INTERVENTIONS:
Drug: Paclitaxel and Carboplatin regimen — Chemotherapy regimen:Paclitaxel: 175mg/m2, d1; Intravenous drip injection with 500ml N.S；Carboplatin: AUC=5, d1; Intravenous drip injection with 500ml G.S Paclitaxel injection at first, followed with Carboplatin injection.
  Other Names: treatment group

SUMMARY:
By detecting the blood concentration of paclitaxel (PTX), Investigator assume this research can identify the individual differences of PTX pharmacokinetics (PK) parameters (TC>0.05 refers to the duration of paclitaxel plasma concentration above 0.05 µmol/L) in Chinese non-small cell lung cancer (NSCLC) patients, and find the correlation between PK results and PTX toxicities and Effectiveness, acquire the optimization method of PTX, and finally try to explore the individualized PTX pharmacokinetically-guided dosing strategy. Orally administer rosiglitazone, which is a substrate of CYP2C8 the same as paclitaxel, before chemotherapy injection. Detect the blood concentration of rosiglitazone, analyze the correlation of rosiglitazone pharmacokinetic parameter and paclitaxel exposure, and explore the effect of rosiglitazone as an in vivo probe of paclitaxel exposure.

1. The variability of paclitaxel concentrations in the patient population dosed by body surface area (BSA), and the limitation of BSA-based dosing of paclitaxel.
2. Verify that paclitaxel TC>0.05 is the most relevant predictor of haematological toxicity and clinical outcomes.
3. Define a dosing algorithm based on paclitaxel TC>0.05 of paclitaxel and quantify its effect on both reducing toxicity and improving Effectiveness.
4. The effect of using dose modification and administration of G-CSF based on toxicity determined by paclitaxel TC>0.05 measurement.
5. Construct a trial outline with the aim of reducing grade 4 neutropenia toxicity and ensuring the clinical outcome by using individual dose adjustments based on the dosing algorithm.
6. Detect the blood concentration of rosiglitazone after orally administration, explore the effect of rosiglitazone as an in vivo probe of paclitaxel exposure based on CYP2C8 activity. Attempt to establish a model to predict the paclitaxel exposure of patients base on rosiglitazone blood concentration before chemotherapy.

DETAILED DESCRIPTION:
Rosiglitazone probe:

Rosiglitazone: time point - at least 20 hours before the initiation of chemotherapy, orally administrate 2mg rosiglitazone.

Only before the first cycle chemotherapy.

Chemotherapy regimen:

Paclitaxel: 175mg/m2, d1; Intravenous drip injection with 500ml N.S Carboplatin: AUC=5, d1; Intravenous drip injection with 500ml G.S Paclitaxel injection at first, followed with Carboplatin injection. 21 days per cycle; 6 cycles in total.

Blood samples collection design:

1. Rosiglitazone blood sample:

   Only one blood sample before 1st cycle:

   - Sample collected 3 hours after orally administration of rosiglitazone, with EDTA blood tube, at least 4ml;
2. Paclitaxel blood samples:

Two blood samples per cycle:

* Sample collected before PTX, with EDTA blood tube, at least 2ml;
* Sample collected 24 hours after the initiation of PTX, with EDTA blood tube, at least 2ml;

Primary Objective:

Object response rate (ORR): assess the ORR of paclitaxel/carboplatin chemotherapy according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1, and analyze the relationship of paclitaxel TC>0.05 and ORR.

Secondary Objectives:

Pharmacokinetic parameters: detect the blood concentration of paclitaxel 24 hours after the initiation, and the blood concentration of rosiglitazone 3 hours after orally administration of rosiglitazone. Calculate paclitaxel TC>0.05 and analyze the correlation of rosiglitazone concentration and paclitaxel TC>0.05.

Toxicities rate: assess the toxicities rate and severity of paclitaxel/carboplatin chemotherapy according to Common Terminology Criteria For Adverse Events (CTCAE) v4.03, and analyze the relationship of paclitaxel TC>0.05 and toxicities.

Survival Effectiveness: assess the progression free survival (PFS) and overall survival (OS) of paclitaxel/carboplatin chemotherapy, analyze the relationship of paclitaxel TC>0.05 and survival Effectiveness.

A single arm, phase II, monocentric, clinical experience trial. The eligible patients sign a informed consent form, and receive a 4 - 6 cycles of paclitaxel/carboplatin chemotherapy. Objective response rate is evaluated by imaging examination (CT or MR scan) every 2 cycles. Toxicities are evaluated by patients' diary for toxicity reports and physician's evaluation at day 10 and day 21 at every cycle. Blood samples are collected every cycle. And survival information is collected by clinic and telephone follow-up.

Response follow-up: An imaging examination should be performed in 4weeks before treatment initiation, and patients are going to receive (CT or MR scan) every 2 cycles during the treatment, the methods should be identical with baseline.

Toxicities follow-up: record the toxicities incident and grades from the first cycle to last cycle until the toxicities relieve or stabilize.

Survival follow-up: after treatment discontinuation, PFS is recorded by imaging examination every 2 cycles (8 weeks) until tumor progression, other anti-cancer treatment start, trial ends or death. OS is recorded by clinic follow-up or telephone follow-up until death.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 ~75 years
* Pathology: Confirmed by pathology (histology or cytology) for advanced non-small cell lung cancer
* Have indications of paclitaxel/carboplatin chemotherapy, suitable for paclitaxel chemotherapy (independent of clinical tumor stage or chemotherapy type or palliative chemotherapy lines)
* At least one measurable tumor lesions (according to RECIST 1.1 criteria)
* ECOG PS score: 0 to 2 points
* Life expectancy: more than 3 months
* Bone marrow reserve function is good, the function of organs (liver and kidney) is good, can satisfy the conditions of implementation chemotherapy. neutrophil count ≥1.5×109/l, platelet ≥75×109/l, hemoglobin >9g/dl, Total Bilirubin ≤1.5×ULN*, transaminase <2.5×ULN*, creatinine ≤1.5×ULN*,or creatinine clearance rate ≥45ml/min. ULR: Upper Limit Of Normal.
* Sign the informed consent form; Compliance is good, can be followed up, willing to comply with the requirements of the study

Exclusion Criteria:

* ECOG Performance Scores > 2 points
* Organic disease (heart, liver, kidney disease etc), Active infection Organ transplantation immunosuppressive therapy, not capable to complete 4 - 6 cycles of paclitaxel / carboplatin chemotherapy.
* Any other tumor history not cured in 3 years before this trial.
* Bone marrow function or organs function not eligible for chemotherapy.
* Diabetic patients currently receiving the standard anti- diabetes treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-03; Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Change of tumor sizes from baseline | baseline; 6 weeks; 12 weeks; 18 weeks; 24 weeks; 32 weeks; up to 3 years.
  Object response rate (ORR): assess the ORR of paclitaxel/carboplatin chemotherapy according to Response Evaluation Criteria In Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of rosiglitazone | 3 hours after rosiglitazone administration
  Detect the plasma concentration of rosiglitazone 3 hours after orally administration of rosiglitazone.
The duration of paclitaxel plasma concentration above 0.05 µmol/L (TC>0.05) | 5min before paclitaxel administration; and 24 hours after.
  Detect the blood concentration of paclitaxel 24 hours after the initiation, Calculate paclitaxel TC>0.05
Toxicities rate | day10, day21, day 31, day 42, day 52, day 63, day 73, day 84, day 94, day 105, day115 and day 126.
  Toxicities rate: assess the toxicities rate and severity of paclitaxel/carboplatin chemotherapy according to Common Terminology Criteria For Adverse Events (CTCAE) v4.03, and analyze the relationship of paclitaxel TC>0.05 and toxicities.
progression free survival (months) | From date of consent form until the date of first documented progression, up to 36 months.
  Survival Effectiveness: assess the progression free survival (PFS) of paclitaxel/carboplatin chemotherapy
Overall survival (months) | From date of consent form until the date of death from any cause, up to 36 months.
  Survival Effectiveness: assess the overall survival (OS) of paclitaxel/carboplatin chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huizing MT, Keung AC, Rosing H, van der Kuij V, ten Bokkel Huinink WW, Mandjes IM, Dubbelman AC, Pinedo HM, Beijnen JH. Pharmacokinetics of paclitaxel and metabolites in a randomized comparative study in platinum-pretreated ovarian cancer patients. J Clin Oncol. 1993 Nov;11(11):2127-35. doi: 10.1200/JCO.1993.11.11.2127. PMID 7901342
- [Background] Kumar N. Taxol-induced polymerization of purified tubulin. Mechanism of action. J Biol Chem. 1981 Oct 25;256(20):10435-41. PMID 6116707
- [Background] Sarosy G, Reed E. Taxol dose intensification and its clinical implications. J Natl Med Assoc. 1993 Jun;85(6):427-31. PMID 8103561
- [Background] Huizing MT, Giaccone G, van Warmerdam LJ, Rosing H, Bakker PJ, Vermorken JB, Postmus PE, van Zandwijk N, Koolen MG, ten Bokkel Huinink WW, van der Vijgh WJ, Bierhorst FJ, Lai A, Dalesio O, Pinedo HM, Veenhof CH, Beijnen JH. Pharmacokinetics of paclitaxel and carboplatin in a dose-escalating and dose-sequencing study in patients with non-small-cell lung cancer. The European Cancer Centre. J Clin Oncol. 1997 Jan;15(1):317-29. doi: 10.1200/JCO.1997.15.1.317. PMID 8996159
- [Background] Joerger M, Huitema AD, Richel DJ, Dittrich C, Pavlidis N, Briasoulis E, Vermorken JB, Strocchi E, Martoni A, Sorio R, Sleeboom HP, Izquierdo MA, Jodrell DI, Calvert H, Boddy AV, Hollema H, Fety R, Van der Vijgh WJ, Hempel G, Chatelut E, Karlsson M, Wilkins J, Tranchand B, Schrijvers AH, Twelves C, Beijnen JH, Schellens JH. Population pharmacokinetics and pharmacodynamics of paclitaxel and carboplatin in ovarian cancer patients: a study by the European organization for research and treatment of cancer-pharmacology and molecular mechanisms group and new drug development group. Clin Cancer Res. 2007 Nov 1;13(21):6410-8. doi: 10.1158/1078-0432.CCR-07-0064. PMID 17975154
- [Background] Miller AA, Rosner GL, Egorin MJ, Hollis D, Lichtman SM, Ratain MJ. Prospective evaluation of body surface area as a determinant of paclitaxel pharmacokinetics and pharmacodynamics in women with solid tumors: Cancer and Leukemia Group B Study 9763. Clin Cancer Res. 2004 Dec 15;10(24):8325-31. doi: 10.1158/1078-0432.CCR-04-1078. PMID 15623609
- [Background] Gianni L, Kearns CM, Giani A, Capri G, Vigano L, Lacatelli A, Bonadonna G, Egorin MJ. Nonlinear pharmacokinetics and metabolism of paclitaxel and its pharmacokinetic/pharmacodynamic relationships in humans. J Clin Oncol. 1995 Jan;13(1):180-90. doi: 10.1200/JCO.1995.13.1.180. PMID 7799018
- [Background] Nakajima M, Fujiki Y, Kyo S, Kanaya T, Nakamura M, Maida Y, Tanaka M, Inoue M, Yokoi T. Pharmacokinetics of paclitaxel in ovarian cancer patients and genetic polymorphisms of CYP2C8, CYP3A4, and MDR1. J Clin Pharmacol. 2005 Jun;45(6):674-82. doi: 10.1177/0091270005276204. PMID 15901749
- [Background] Mould DR, Fleming GF, Darcy KM, Spriggs D. Population analysis of a 24-h paclitaxel infusion in advanced endometrial cancer: a gynaecological oncology group study. Br J Clin Pharmacol. 2006 Jul;62(1):56-70. doi: 10.1111/j.1365-2125.2006.02718.x. PMID 16842379
- [Background] Kobayashi M, Oba K, Sakamoto J, Kondo K, Nagata N, Okabayashi T, Namikawa T, Hanazaki K. Pharmacokinetic study of weekly administration dose of paclitaxel in patients with advanced or recurrent gastric cancer in Japan. Gastric Cancer. 2007;10(1):52-7. doi: 10.1007/s10120-006-0411-6. Epub 2007 Feb 23. PMID 17334719
- [Background] Jiko M, Yano I, Sato E, Takahashi K, Motohashi H, Masuda S, Okuda M, Ito N, Nakamura E, Segawa T, Kamoto T, Ogawa O, Inui K. Pharmacokinetics and pharmacodynamics of paclitaxel with carboplatin or gemcitabine, and effects of CYP3A5 and MDR1 polymorphisms in patients with urogenital cancers. Int J Clin Oncol. 2007 Aug;12(4):284-90. doi: 10.1007/s10147-007-0681-y. Epub 2007 Aug 20. PMID 17701008
- [Background] Ohtsu T, Sasaki Y, Tamura T, Miyata Y, Nakanomyo H, Nishiwaki Y, Saijo N. Clinical pharmacokinetics and pharmacodynamics of paclitaxel: a 3-hour infusion versus a 24-hour infusion. Clin Cancer Res. 1995 Jun;1(6):599-606. PMID 9816021
- [Background] Spratlin J, Sawyer MB. Pharmacogenetics of paclitaxel metabolism. Crit Rev Oncol Hematol. 2007 Mar;61(3):222-9. doi: 10.1016/j.critrevonc.2006.09.006. Epub 2006 Nov 7. PMID 17092739
- [Background] Mielke S, Sparreboom A, Steinberg SM, Gelderblom H, Unger C, Behringer D, Mross K. Association of Paclitaxel pharmacokinetics with the development of peripheral neuropathy in patients with advanced cancer. Clin Cancer Res. 2005 Jul 1;11(13):4843-50. doi: 10.1158/1078-0432.CCR-05-0298. PMID 16000582
- [Background] Augusto C, Pietro M, Cinzia M, Sergio C, Sara C, Luca G, Scaioli V. Peripheral neuropathy due to paclitaxel: study of the temporal relationships between the therapeutic schedule and the clinical quantitative score (QST) and comparison with neurophysiological findings. J Neurooncol. 2008 Jan;86(1):89-99. doi: 10.1007/s11060-007-9438-8. Epub 2007 Jul 5. PMID 17611715
- [Background] Dai D, Zeldin DC, Blaisdell JA, Chanas B, Coulter SJ, Ghanayem BI, Goldstein JA. Polymorphisms in human CYP2C8 decrease metabolism of the anticancer drug paclitaxel and arachidonic acid. Pharmacogenetics. 2001 Oct;11(7):597-607. doi: 10.1097/00008571-200110000-00006. PMID 11668219
- [Background] Mielke S, Sparreboom A, Behringer D, Mross K. Paclitaxel pharmacokinetics and response to chemotherapy in patients with advanced cancer treated with a weekly regimen. Anticancer Res. 2005 Nov-Dec;25(6C):4423-7. PMID 16334120
- [Background] Joerger M, Huitema AD, van den Bongard DH, Schellens JH, Beijnen JH. Quantitative effect of gender, age, liver function, and body size on the population pharmacokinetics of Paclitaxel in patients with solid tumors. Clin Cancer Res. 2006 Apr 1;12(7 Pt 1):2150-7. doi: 10.1158/1078-0432.CCR-05-2069. PMID 16609028
- [Background] Hertz DL, Walko CM, Bridges AS, Hull JH, Herendeen J, Rollins K, Watkins PB, Dees EC. Pilot study of rosiglitazone as an in vivo probe of paclitaxel exposure. Br J Clin Pharmacol. 2012 Jul;74(1):197-200. doi: 10.1111/j.1365-2125.2012.04165.x. PMID 22680343
- [Background] Frye RF. Probing the world of cytochrome P450 enzymes. Mol Interv. 2004 Jun;4(3):157-62. doi: 10.1124/mi.4.3.5. PMID 15210869
- [Background] Sparreboom A, Huizing MT, Boesen JJ, Nooijen WJ, van Tellingen O, Beijnen JH. Isolation, purification, and biological activity of mono- and dihydroxylated paclitaxel metabolites from human feces. Cancer Chemother Pharmacol. 1995;36(4):299-304. doi: 10.1007/BF00689047. PMID 7628049
- [Background] Freed MI, Allen A, Jorkasky DK, DiCicco RA. Systemic exposure to rosiglitazone is unaltered by food. Eur J Clin Pharmacol. 1999 Mar;55(1):53-6. doi: 10.1007/s002280050592. PMID 10206085
- [Background] Baldwin SJ, Clarke SE, Chenery RJ. Characterization of the cytochrome P450 enzymes involved in the in vitro metabolism of rosiglitazone. Br J Clin Pharmacol. 1999 Sep;48(3):424-32. doi: 10.1046/j.1365-2125.1999.00030.x. PMID 10510156
- [Background] Naik H, Wu JT, Palmer R, McLean L. The effects of febuxostat on the pharmacokinetic parameters of rosiglitazone, a CYP2C8 substrate. Br J Clin Pharmacol. 2012 Aug;74(2):327-35. doi: 10.1111/j.1365-2125.2012.04182.x. PMID 22242967
- [Background] Bjornsson TD, Callaghan JT, Einolf HJ, Fischer V, Gan L, Grimm S, Kao J, King SP, Miwa G, Ni L, Kumar G, McLeod J, Obach SR, Roberts S, Roe A, Shah A, Snikeris F, Sullivan JT, Tweedie D, Vega JM, Walsh J, Wrighton SA; Pharmaceutical Research and Manufacturers of America Drug Metabolism/Clinical Pharmacology Technical Working Groups. The conduct of in vitro and in vivo drug-drug interaction studies: a PhRMA perspective. J Clin Pharmacol. 2003 May;43(5):443-69. PMID 12751267
- [Background] Sahi J, Black CB, Hamilton GA, Zheng X, Jolley S, Rose KA, Gilbert D, LeCluyse EL, Sinz MW. Comparative effects of thiazolidinediones on in vitro P450 enzyme induction and inhibition. Drug Metab Dispos. 2003 Apr;31(4):439-46. doi: 10.1124/dmd.31.4.439. PMID 12642470
- [Background] Joerger M, Kraff S, Huitema AD, Feiss G, Moritz B, Schellens JH, Beijnen JH, Jaehde U. Evaluation of a pharmacology-driven dosing algorithm of 3-weekly paclitaxel using therapeutic drug monitoring: a pharmacokinetic-pharmacodynamic simulation study. Clin Pharmacokinet. 2012 Sep 1;51(9):607-17. doi: 10.1007/BF03261934. PMID 22804749